CLINICAL TRIAL: NCT03354780
Title: Impact of Endometriosis on the Risk of Miscarriage in Spontaneous Pregnancy: a Multicentric Italian Study
Brief Title: Endometriosis and Risk of Miscarriage
Status: Completed | Type: Observational
Sponsor: Endometriosis Treatment Italian Club (Other)
Collaborators: University of Milan (Other)
Responsible Party: Sponsor
Other Study IDs: ETIC001
Record Dates: First submitted 2017-11-21; First posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Endometriosis; Miscarriage
MeSH Terms: conditions — Endometriosis; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- endometriosis: Survey on first pregnancy after endometriosis diagnosis
  Interventions: Other: Survey on first pregnancy after endometriosis diagnosis
- non endometriosis: Survey on first pregnancy
  Interventions: Other: Survey on first pregnancy

INTERVENTIONS:
Other: Survey on first pregnancy after endometriosis diagnosis — rate of miscarriage was noted
  Groups: endometriosis
Other: Survey on first pregnancy — rate of miscarriage was noted
  Groups: non endometriosis

SUMMARY:
The aim of this study is to compare the rate of miscarriage at first spontaneous pregnancy among women with endometriosis with the rate of miscarriage at first spontaneous pregnancy among women without endometriosis.

DETAILED DESCRIPTION:
All women followed up for a surgical or sonographic diagnosis of endometriosis in 11 italian referral Centres for the treatment of endometriosis completed a questionnaire regarding their previous pregnancies. The same questionnaire was completed by women, attending a routine gynecologic visit, in whom surgery or vaginal examination and pelvic ultrasonography excluded endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* 30 to 50 years old women
* with at least one previous spontaneous pregnancy
* with surgical or clinical/sonographic diagnosis of endometriosis or
* in whom surgical or clinical/sonographic evaluation ruled out endometriosis

Exclusion Criteria:

* Pregnancy achieved by Assisted Reproductive technology
* Biochemical pregnancy
* Non corrected uterine malformation, poliabortivity, lupus like anticoagulant

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: All continous women attending endometriosis clinics or undergoing a routine gynecological examination matching the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 844 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2017-10-04 (Actual)

PRIMARY OUTCOMES:
Rate of miscarriage | 2 years
  comparison of rate of miscarriage in the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Berlanda, MD, Principal Investigator — Endometriosis Treatment Italian Club